CLINICAL TRIAL: NCT05673031
Title: 68Ga-HA-DOTATATE PET/CT in Adults With Neuroendocrine Tumors
Status: Recruiting | Type: Observational
Sponsor: Alberta Health services (Other)
Responsible Party: Principal Investigator, Dr. Denise Chan, Clinical Assistant Professor, Alberta Health services
Other Study IDs: NM-CRS-002
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Neuroendocrine Tumors (NET)
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 68Ga-HA-DOTATATE: 68Ga-HA-DOTATATE Intravenous injection of 100-250 MBq 68Ga-HA-DOTATATE
  Interventions: Diagnostic Test: 68Ga-HA-DOTATATE PET/CT imaging

INTERVENTIONS:
Diagnostic Test: 68Ga-HA-DOTATATE PET/CT imaging — Each patient will receive an IV injection 68Ga-HA-DOTATATE. Imaging will be conducted beginning 45-90 minutes after an injection of between 100-250 MBq 68Ga-HA-DOTATATE in patients.
  * After the 68Ga-HA-DOTATATE acquisition is complete, a CT scan will be performed for attenuation correction and localization in the same in line gantry without patient movement between the two scans.
  * The results of the 68Ga-HA-DOTATATE PET/CT will be compared to any prior imaging and pathologic results.

SUMMARY:
To determine if 68Ga-HA-DOTATATE PET/CT imaging is effective at diagnosing somatostatin positive tumors compared to conventional imaging [including CT, MRI, 111 In-pentetreotide Scans, 18F-FDG PET/CT, as available]

DETAILED DESCRIPTION:
The purpose of the current study will be to evaluate the usefulness of 68Ga-HA-DOTATATE compared to current standard anatomical imaging including CT, MRI, 111 In-pentetreotide Scans, 18F-FDG PET/CT, as available. Specifically, we aim to assess the utility of 68Ga-HA-DOTATATE in primary workup of neuroendocrine tumours, including suspected neuroendocrine tumours that do not have a cross-sectional imaging correlate. An additional aim is to assess the role of 68Ga-HA-DOTATATE in surveillance of completely resected neuroendocrine tumours, which is a point of disagreement amongst current society guidelines . Finally, we will assess utility of 68Ga-HA-DOTATATE for localization of functioning neuroendocrine tumors including insulinoma and gastrinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female. If female of child-bearing potential and outside of the window of 10 days since the last menstrual period, a negative pregnancy test will be required.
2. Age greater than or equal to 18 years.
3. Able and willing to follow instructions and comply with the protocol.
4. Provide written informed consent prior to participation in the study.
5. Clinically suspected (patients presenting with symptom(s) suggestive of carcinoid syndrome or biochemically suggestive of Neuroendocrine Tumor) or Biopsy proven Neuroendocrine Tumor

Exclusion Criteria:

1. Nursing or pregnant females.
2. Age less than 18 years.
3. Surgery in the area of interest within the preceding 2 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically suspected (patients presenting with symptom(s) suggestive of carcinoid syndrome or biochemically suggestive of Neuroendocrine Tumor) or Biopsy proven Neuroendocrine Tumor. Patients greater than 18 years of age who are able to follow instructions and provide written consent to participate in study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
68Ga-HA-DOTATATE PET/CT imaging | 5 years
  To compare 68Ga-HA-DOTATATE PET/CT imaging at identifying somatostatin positive tumors to conventional imaging [including CT, MRI, 111 In-pentetreotide Scans, 18F-FDG PET/CT, as available]. 68Ga-HA-DOTATATE PET/CT scans will be evaluated for abnormal accumulation of 68Ga-HA-DOTATATE. Any abnormal uptake will be determined for up to 5 lesions and compared to results of standard of care imaging performed [including CT, MRI, 111 In-pentetreotide (OctreoscanTM) Scan with SPECT/CT, 18F-FDG PET/CT, as available] for presence/absence of each lesion. Comparison to any follow up 68Ga-HA-DOTATATE PET/CT Scans will also be performed (up to 5 follow up68Ga-HA-DOTATATE PET/CT Scans will be allowed).

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Center 1403 29 St NW, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No